CLINICAL TRIAL: NCT06973525
Title: Optimizing Neoadjuvant Therapy for HER2-Positive Breast Cancer Based on Dynamic Efficacy Monitoring: A Trial of Trastuzumab Plus Pyrotinib and Albumin-Bound Paclitaxel Followed by SHR-A1811 Plus Pertuzumab（OnThePath Trial）
Brief Title: This Study Aims to Optimize Neoadjuvant Therapy for HER2-positive Breast Cancer by Implementing a Dynamic Monitoring-guided Treatment Strategy.
Acronym: HER2-DM-NACT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pending Assignment
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811+Pertuzumab (Experimental): Patients will initially receive trastuzumab, pyrotinib, and albumin-bound paclitaxel. Those who do not achieve a radiological response after Cycle 2 will switch to SHR-A1811 (a HER2-targeted antibody-drug conjugate) combined with pertuzumab.
  Interventions: Drug: Patients will initially receive trastuzumab, pyrotinib, and albumin-bound paclitaxel. Those who do not achieve a radiological response after Cycle 2 will switch to SHR-A1811 (a HER2-targeted antibody
- trastuzumab, pyrotinib, and nab-paclitaxe (Active Comparator): Patients will initially receive trastuzumab, pyrotinib, and nab-paclitaxel. Those who achieve a partial response (PR) or complete response (CR) after cycle 2 will continue on the same regimen.
  Interventions: Drug: Patients will initially receive trastuzumab, pyrotinib, and nab-paclitaxel. Those who achieve a partial response (PR) or complete response (CR) after cycle 2 will continue on the same regimen.

INTERVENTIONS:
Drug: Patients will initially receive trastuzumab, pyrotinib, and albumin-bound paclitaxel. Those who do not achieve a radiological response after Cycle 2 will switch to SHR-A1811 (a HER2-targeted antibody — Drug: SHR-A1811 Drug: Pertuzumab
  Arms: SHR-A1811+Pertuzumab
Drug: Patients will initially receive trastuzumab, pyrotinib, and nab-paclitaxel. Those who achieve a partial response (PR) or complete response (CR) after cycle 2 will continue on the same regimen. — Patients will initially receive trastuzumab, pyrotinib, and nab-paclitaxel. Those who achieve a partial response (PR) or complete response (CR) after cycle 2 will continue on the same regimen.
  Arms: trastuzumab, pyrotinib, and nab-paclitaxe

SUMMARY:
This study aims to optimize neoadjuvant therapy for HER2-positive breast cancer by implementing a dynamic monitoring-guided treatment strategy. Patients will initially receive trastuzumab, pyrotinib, and albumin-bound paclitaxel. Those who do not achieve a radiological response after Cycle 2 will switch to SHR-A1811 (a HER2-targeted antibody-drug conjugate) combined with pertuzumab. The primary objective is to evaluate whether this sequential treatment strategy improves the pathological complete response (pCR) rate while maintaining safety. The study will also explore the value of dynamic efficacy monitoring in guiding treatment adjustments and assess the safety and tolerability of the regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive cancer of the breast and meet the clinical stage II（T2N0-1M0/T3N0M0）or III（T2N2M0/T3N1-2M0) criteria;
2. Age between18-70 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
4. Histologically confirmed to be HER2-positive invasive breast cancer;
5. LVEF≥55%；
6. At least one measurable lesion according to RECIST version 1.1
7. Normal organ and marrow function: Hemoglobin (HB) ≥90 g/L (No blood was transfused within 14 days), Absolute neutrophil count ≥ 1500/μL, Platelets ≥ 75,000/μL, Total bilirubin ≤ 1.5 x ULN), aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 3 x ULN, creatinine < 1 x ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
8. Non-pregnant and non-lactating, fertile female subjects were required to use a medically approved contraceptive method for the duration of the study treatment and at least 3 months after the last use of the study drug; Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer.
2. The patient has a second primary malignant tumor, except for fully treated skin cancer.
3. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or the patient has not fully recovered from such surgical procedures.
4. The presence of uncontrolled cardiovascular and cerebrovascular disease, including (but not limited to) any of the following within the 6 months prior to the first dose: congestive heart failure (NYHA III or IV), myocardial infarction or cerebral infarction, pulmonary embolism, unstable angina, or arrhythmia requiring treatment at the time of screening; 5.Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restricted cardiomyopathy, undefined cardiomyopathy); A clinically significant history of prolonged QTc, grade II type II atrioventricular block or grade III atrioventricular block or QTc interphase (F method) > 470 msec (female); Atrial fibrillation (EHRA grade ≥2b); Unmanageable hypertension, which the investigators judged unsuitable for study participation.

6.Individuals with a known history of allergies to the drug components of this protocol; 7.Having a history of immunodeficiency, including HIV testing positive, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
tpCR | At the time of surgery
  Total pathological complete response (tpCR: ypT0-is/ypN0)

SECONDARY OUTCOMES:
EFS | 5 years
  Event-free survival

OTHER OUTCOMES:
bpCR | At the time of surgery
  Breast pathological complete response (bpCR：ypT0-is)
ORR | During 24 weeks of the neoadjuvant treatment
  Objective Response Rate (ORR) according to Response Evaluation Criteria in Solid
Incidence of Adverse Events | from consent to 28 days after last dose
  Incidence of Adverse Events

IPD SHARING:
Plan to Share IPD: No